CLINICAL TRIAL: NCT05095077
Title: Effects of Single Dose Tadalafil on Urethral and Anal Closure Function and on Urinary Flow in Healthy Females: A Randomised, Controlled, Double-blinded, Two-period Cross-over Study
Brief Title: Effects of Single Dose Tadalafil on Urethral and Anal Closure Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Thea Christoffersen, Medical Doctor, Principal Investigator, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PDE5I-UPR-AAR-01; 2020-005839-76 (EudraCT Number)
Record Dates: First submitted 2021-08-26; First posted 2021-10-27 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Urinary Incontinence,Stress; Fecal Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Fecal Incontinence | interventions — Tadalafil

STUDY DESIGN:
Intervention Model Description: Two-period (AB/BA) crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The tadalafil tablets and placebo are over-encapsulated in identical hard-gelatin capsules. The over-encapsulation, packaging and labelling is performed by the hospital pharmacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tadalafil (Experimental): Subjects are randomized to either 40 mg tadalafil on study day 1 and placebo on study day 2, or placebo on study day 1 and 40 mg tadalafil on study day 2.
  Interventions: Drug: Tadalafil 40 MG
- Placebo (Placebo Comparator): Subjects are randomized to either 40 mg tadalafil on study day 1 and placebo on study day 2, or placebo on study day 1 and 40 mg tadalafil on study day 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil 40 MG — Single dose on study day 1/2
  Arms: Tadalafil
Drug: Placebo — Identical to active IMP
  Arms: Placebo

SUMMARY:
The purpose of the trial is to assess the effect of tadalafil compared to placebo (inactive comparator) on the urethral - and anal pressure and on urine flow in healthy females. Further, the purpose of the trial is to evaluate the potential for going forward with studies of tadalafil in patients suffering from urine or fecal incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Normal weight (Body weight 50 kg or more, Body Mass Index 18-5-30 kg/m2)
* Sexual abstinence or use of safe contraceptive methods i.e. intrauterine devices, hormonal contraception (oral contraceptive pills, implants, transdermal patches, vaginal rings or long acting injections), or surgically sterilized partner throughout the course of the study and until six days after the study has ended for the subject. Women who are postmenopausal (defined as no menstrual periods for 12 months or more prior to enrolment) can be included without use of contraceptive methods.
* Presentation of a negative urine human chorionic gonadotropin (hCG) urine pregnancy test prior to dosing (on both study days)

Exclusion Criteria:

* History of clinically significant urinary incontinence.
* Current acute or chronic condition, unless considered clinically irrelevant and stable by the investigator.
* Average systolic blood pressure <100 mmHg or >140 mmHg and/or average diastolic blood pressure <60 mmHg or >90 mmHg (average of three measurements performed at screening).
* Average pulse < 40 or > 100 beats/minute (average of three measurements performed at screening).
* Pregnancy within 6 months before screening and throughout the study period.
* Breastfeeding throughout the study period and 6 days after study day 2.
* Any systemic drug use within 2 weeks before first study drug administration (prescription drugs, over-the-counter drugs, herbal drugs and illicit drugs), except for occasional use of paracetamol (up to 4 g/day), hormonal contraceptives and hormone replacement therapy.
* Smoking or other regular use of any form of nicotine product during the study period and the previous 3 months.
* Alcohol consume 24 hours prior to dosing.
* Current or prior participation (within 3 months before screening) in other clinical trials that might affect the results of this study (judged by the investigator).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected change in opening urethral pressure after single dose tadalafil | 2 hours post-dose
  Difference in average urethral opening pressure (UOP) after administration of 40 mg tadalafil (UOP-tadalafil) compared to UOP after placebo (during relaxation).

SECONDARY OUTCOMES:
Difference in average anal opening pressure (AOP) after administration of 40 mg tadalafil compared to AOP after placebo (during relaxation). | 2-hours post-dose
  Difference in average anal opening pressure (AOP) after administration of 40 mg tadalafil compared to AOP after placebo (during relaxation).
Difference in average UOP-tadalafil and average UOP-placebo during squeezing. | 2-hours post-dose
Difference in average AOP-tadalafil and average AOP-placebo during squeezing. | 2-hours post-dose
Elastance (opening/closing) during relaxation and squeezing (tadalafil compared to placebo). | 2-hours post-dose
Difference in maximum urine flow rate (Qmax) and average urine flow rate (Qave) after tadalafil and placebo administration, respectively. | 2-hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Thea Christoffersen, Principal Investigator — Zelo Phase 1 unit, University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Zelo Phase 1 unit, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided